CLINICAL TRIAL: NCT06030830
Title: SMaRT Mom - Smartphone Management and Responsive Time for Breastfeeding Mothers - An Intervention Study
Brief Title: SMaRT Mom - Smartphone Management and Responsive Time for Breastfeeding Mothers
Acronym: SMaRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Prof. Ilanit gordon, prof., Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IG30623
Record Dates: First submitted 2023-08-27; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Smartphone Addiction; Breastfeeding; Infant Behavior; Mother-Infant Interaction
Keywords: Smartphone addiction; Problematic smartphone use; Breastfeeding; Infant temperament; Mother-infant interaction
MeSH Terms: conditions — Internet Addiction Disorder; Breast Feeding; Infant Behavior

STUDY DESIGN:
Intervention Model Description: The SMaRT Mom intervention plan will be administered for one week during which mothers will be instructed not using their smartphone while breastfeeding. Before and after the intervention week, two lab sessions will be take place in which mothers in both intervention and control groups will be asked to take a screen shot of their smart digital use of the past week, and will be connected to the electrophysiological monitoring systems to assess their biobehavioral responses during: baseline, the smartphone cue-reactivity task, breastfeeding and face-to-face interaction while using or not using the smartphone. Following the first lab visit, mothers will be instructed to follow the intervention program. The participants will be asked to complete three daily reports of any distractions while breastfeeding. During the intervention week, two remote sessions (20 minutes each) will be performed by a research assistance to support the implementation of the intervention plan.
Who Masked: Participant
Masking Description: The intervention given to the intervention group will be hidden from participants in the control group, and they will not be asked to refrain from using their smartphones for a week. Participants in the control group will be given information about the intervention week after the second lab visit and allowed to undergo the same intervention the following week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be instructed not to use the smartphone during breastfeeding for a week
  Interventions: Behavioral: SMaRT Mom
- Control (No Intervention): Participants will not be instructed not to use the smartphone during breastfeeding for a week

INTERVENTIONS:
Behavioral: SMaRT Mom — "SMaRT Mom" intervention that we have developed is based on several approaches to digital addiction detection, prevention, and intervention aimed to help breastfeeding mothers to manage and reduce smartphone use during breastfeeding. The SMaRT Mom intervention results will be measured in changes in two main outcomes: 1) reduced maternal reports of their infants' negative emotionality, and 2) increased maternal self-efficacy as distal outcomes as well as two proximal outcomes: 1) breastfeeding as a rewarding experience, and 2) maternal attention towards their infant during breastfeeding. We will then assess changes in breastfeeding mothers' neural activity, physiology and behavior before and after the implementation of the SMaRT Mom intervention, as potential mechanisms underlying changes in the main outcomes of the intervention.
  Arms: Intervention

SUMMARY:
In the last decade, infants are born into a social environment in which the smartphone has become an essential part of our lives. Smartphone use draws the mother's attention during mother-infant interactions and thus may affect the infant development as well as maternal self-efficacy. However, the effects of smartphone use reduction among breastfeeding mothers during their interactions with their infants have not been studied yet. In the present study, we propose to evaluate a "SMaRT Mom" intervention that we have developed, to manage and reduce smartphone use during breastfeeding. The purpose of the study is to evaluate the effects of the SMaRT Mom intervention on breastfeeding mothers' biobehavioral mechanisms, self-efficacy and the socioemotional characteristics of their infants. This will extend our knowledge of the peculiarities of early mother-infant interactions in the digital era, when smartphones play a critical role.

ELIGIBILITY:
Inclusion Criteria:

* 3-6 months old infant
* Smartphone Addiction Scale' cut-off (31 and above)

Exclusion Criteria:

* No neurological disorders
* No heart disease
* No anxiety and depression
* No use of psychiatric drugs

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy breastfeeding mothers
Enrollment: 100 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Infant temperament | Pre (day 1) and post (day 8) lab visit (before and after intervention/control week)
  Infants' temperament will be reported by breastfeeding mothers before and after the intervention week using the Infant Behavior Questionnaire - Revised - Very Short Form (IBQ-rvsf). Scale scores represent the mean score of all scale items applicable to the child, as judged by the caregiver. 1. Sum all numerical item responses for a given scale. Note that: a) If caregiver omitted an item, that item receives no numerical score; b) If caregiver checked the "does not apply" response option for an item, that item receives no numerical score; 2. Divide the total by the number of items receiving a numerical response. Not including items marked "does not apply (N/A)" or items receiving no response in determining the number of items. The surgency, negative affect and effortful control subscales' items will be averaged
Maternal self-efficacy | Pre (day 1) and post (day 8) lab visit (before and after intervention/control week)
  Maternal self-efficacy questionnaire (MSQ) will be self-reported by breastfeeding mothers before and after the intervention week.
  The scale applies a special method to measure maternal self-efficacy and mostly focuses on a mother's infant care responsibilities.
  The scale consists of 10 items.Higher score indicates higher maternal self-efficacy

SECONDARY OUTCOMES:
Breastfeeding as a rewarding experience | Pre (day 1) and post (day 8, day 14, day 30) lab visit after intervention/control week
  The rewarding experience of breastfeeding will be self-reported by mothers before and after the intervention week ("How rewarding is the experience of breastfeeding for you?")
Self-reported maternal attention towards infant | Pre (day 1) and post (day 8, day 14, day 30) lab visit after intervention/control week
  Maternal attention towards the infant will be self-reported by mothers before and after the intervention week ("How attentive do you feel towards your infant during breastfeeding?")
Video recorded maternal attention towards infant | day 1 and day 8 during lab visits
  Maternal attention towards the infant will be video recorded during both laboratory sessions
Changes in breastfeeding mothers' neural activity - Frontal asymmetry | day 1 and day 8 during lab visits
  Frontal asymmetry during maternal baseline, breastfeeding and mother-infant face-to-face interaction EEG data will be acquired from breastfeeding mothers' heads using Enobio8 device with eight electrodes from the frontal, and central-parietal areas - Fp1, Fp2, F3, F4, F7, F8, P3 and P4 and voltage fluctuations in the alpha frequency band will be measured between pairs of electrodes that will be produced by the excitation of neuronal synapses.
Changes in breastfeeding mothers' neural activity - ERP | day 1 and day 8 during lab visits
  Event related response during the smartphone cue-reactivity task, attentional bias is indicated by an enhancement in the late positive potential (LPP), which is strongly evoked by emotionally salient stimuli. The LPP is maximum over central-parietal regions occurring between 300 and 700 ms following an emotional stimulus
Changes in breastfeeding mothers' physiological responses - HRV | day 1 and day 8 during lab visits
  Heart Rate Variability (HRV) will be measured via The MindWare Mobile Recorder (MindWare Technologies, Inc., Gahanna, OH), a well-validated and specialized hardware and software system that is aimed at monitoring autonomic balance, cardiac performance, respiratory measurements and activity. Participants are each will be fitted with a MindWare Mobile device and specialized electrodes to measure the electrocardiogram (allows to derive HRV), Z0, dz/dt (allows to assess respiration and cardiology impedance) and SCL (allows to derive electrodermal activity from the skin) (for similar method see Nomkin & Gordon, 2021).
Changes in breastfeeding mothers' physiological responses - Electrodermal activity | day 1 and day 8 during lab visits
  Skin Conductance Level (SCL) will be measured via The MindWare Mobile Recorder (MindWare Technologies, Inc., Gahanna, OH), a well-validated and specialized hardware and software system that is aimed at monitoring autonomic balance, cardiac performance, respiratory measurements and activity. Participants are each will be fitted with a MindWare Mobile device and specialized electrodes to measure the electrocardiogram (allows to derive HRV), Z0, dz/dt (allows to assess respiration and cardiology impedance) and SCL (allows to derive electrodermal activity from the skin) (for similar method see Nomkin & Gordon, 2021).
Changes in breastfeeding mothers' physiological responses - Cardiograph Impedance | day 1 and day 8 during lab visits
  Cardiograph Impedance will be measured via The MindWare Mobile Recorder (MindWare Technologies, Inc., Gahanna, OH), a well-validated and specialized hardware and software system that is aimed at monitoring autonomic balance, cardiac performance, respiratory measurements and activity. Participants are each will be fitted with a MindWare Mobile device and specialized electrodes to measure the electrocardiogram (allows to derive HRV), Z0, dz/dt (allows to assess respiration and cardiology impedance) and SCL (allows to derive electrodermal activity from the skin) (for similar method see Nomkin & Gordon, 2021).

CONTACTS AND LOCATIONS:
Overall Officials: Ilanit Gordon, Prof., Study Chair — Department of Psychology, Gonda Brain Research Center Bar-Ilan University
Locations (1):
- Gonda Brain Center, Bar-Ilan University, Ramat Gan, Israel